CLINICAL TRIAL: NCT06375655
Title: A Proposed Randomized Clinical Trial of the Effectiveness of a New Breastfeeding- Supportive Texting Program Designed Specifically for African-American/Black Expectant Women, as Compared to a National Maternal Health Texting Program, on Rates of Exclusive Breastfeeding at 2 Months
Brief Title: Texting to Promote Breastfeeding (TOPS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY20240085
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Results first posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Increased Breastfeeding
Keywords: African American; Texting; Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Team2BF (Experimental): Team2BF includes 3-4 breastfeeding-supportive messages per time interval, sent weekly from 28 weeks gestation through delivery, daily through 2 weeks postpartum, weekly from 2 to 10 weeks, and then monthly to one year. Other maternal health topics are not addressed.
  Interventions: Behavioral: Team2BF
- Bright By Text (Active Comparator): Bright By Text sends 2-4 messages per week from the first trimester through and beyond one year postpartum about a wide range of maternal and child health topics as outlined on their website; 8 messages are specifically about breastfeeding.
  Interventions: Behavioral: Bright By Text

INTERVENTIONS:
Behavioral: Team2BF — Team2BF includes 3-4 breastfeeding-supportive messages per time interval, sent weekly from 28 weeks gestation through delivery, daily through 2 weeks postpartum, weekly from 2 to 10 weeks, and then monthly to one year. Other maternal health topics are not addressed.
  Arms: Team2BF
Behavioral: Bright By Text — Bright By Text sends 2-4 messages per week from the first trimester through and beyond one year postpartum about a wide range of maternal and child health topics as outlined on their website; 8 messages are specifically about breastfeeding.
  Arms: Bright By Text

SUMMARY:
The purpose of the study is to see if a program of text messages that support and promote breastfeeding for expecting and delivered African-American/Black women (called TEAM2BF), as compared to a national maternal health texting program (called Bright By Text), can result in more women being able to breastfeed their infant. Because breastfeeding is healthy for mothers and babies, and because fewer African-American/Black women decide to breastfeed and continue breastfeeding than many other racial and ethnic groups, researchers like us are trying to figure out ways to be supportive to African-American/Black mothers who might be interested in breastfeeding. The investigators will enroll up to 80 mothers and their infants at UHCMC.

ELIGIBILITY:
Inclusion Criteria:

* Expectant women initiating obstetrical care <34 weeks or at any prenatal visit up to 34 weeks gestation
* Daily access to a mobile phone with text message capabilities,
* Self-identify as African-American/Black,
* English speaking, and
* Infant feeding plan of "might or will breastfeed"
* Receive care at Ahuja Midtown or MAC1200

Exclusion Criteria:

* Committed to feeding formula only to their infant
* No mobile phone with text capability

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 83 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Furman, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Ahuja Rainbow Center for Women and Children, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred in person in obstetrical clinics at the Rainbow Ahuja Women and Children's Center from 7/1/24-11/5/24
Pre-assignment Details: Enrolled participants were not removed from the study prior to assignment. Three participants delivered prematurely and 3 new participants were recruited in their places to achieve 80 total participants.
Period: Overall Study
Arm/Group | Team2BF | Bright By Text
Started | 42 | 41
Completed | 40 | 40
Not Completed | 2 | 1
Not completed — premature delivery (prior to 35 weeks GA) | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Team2BF | Bright By Text | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.68 (5.55) | 25.78 (5.34) | 26.23 (5.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 40 | 40 | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 40 | 40 | 80
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who do Not Opt Out of Receipt of Text Messages
Time Frame: Up to 6 months postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Team2BF | Bright By Text
Number analyzed (Participants) | 40 | 40
Participants | 40 | 40
Statistical Analysis 1: Comparison: Team2BF vs Bright By Text; Test type: Other; p = 1, Fisher Exact; Odds Ratio (OR) = 0

2. Primary Outcome: Number of Participants Who Said Texts Were Helpful as Measured by Questionnaire
Description: Participants were asked if texts were helpful- yes or no. Reported on number of participants who said yes.
Time Frame: Up to 6 months postpartum
Population: Not all participants responded
Measure: Count of Participants; unit: Participants
Arm/Group | Team2BF | Bright By Text
Number analyzed (Participants) | 26 | 27
Participants | 22 | 20
Statistical Analysis 1: Comparison: Team2BF vs Bright By Text; This analysis did not power the study; Test type: Superiority; p = 0.5007, Fisher Exact; Odds Ratio (OR) = 1.901509, 95% CI 2-sided [0.41 to 10.25]

3. Primary Outcome: Number of Participants Who Would Refer a Friend/Family to the Texting Program
Description: This will be a yes/no answer
Time Frame: Up to 6 months postpartum
Population: All participants did not provide a response
Measure: Count of Participants; unit: Participants
Arm/Group | Team2BF | Bright By Text
Number analyzed (Participants) | 26 | 26
Participants | 25 | 22
Statistical Analysis 1: Comparison: Team2BF vs Bright By Text; Test type: Superiority; p = 0.3497, Fisher Exact; Odds Ratio (OR) = 4.43, 95% CI 2-sided [0.3986 to 232.3218]

4. Secondary Outcome: Number of Participants Who Are Exclusively Breastfeeding at 2 Months Postpartum as Measured by Participant Report/Chart Review
Time Frame: Up to 2 months postpartum
Population: Missing information from one participant
Measure: Count of Participants; unit: Participants
Arm/Group | Team2BF | Bright By Text
Number analyzed (Participants) | 39 | 40
Participants | 16 | 18
Statistical Analysis 1: Comparison: Team2BF vs Bright By Text; Test type: Superiority; p = 0.7, Chi-squared

5. Secondary Outcome: Change in the Number of Participants Who Are Exclusively Breastfeeding as Measured by Participant Report/Chart Review
Time Frame: 1 month, 3 months, 6 months postpartum
Population: None missing at 1 month, 1 missing at 3 and 6 months for Team2BF, 0 missing at 3 months and 2 at 6 months for Bright By Text
Measure: Count of Participants; unit: Participants
Arm/Group | Team2BF | Bright By Text
Number analyzed (Participants) | 40 | 40
Participants
  1 month postpartum | 18 | 22
  3 months postpartum: number analyzed (Participants) | 39 | 40
  3 months postpartum | 10 | 15
  6 months postpartum: number analyzed (Participants) | 39 | 38
  6 months postpartum | 7 | 11
Statistical Analysis 1: Comparison: Team2BF vs Bright By Text; Test type: Superiority; p = 0.2302, Cochran-Mantel-Haenszel — Value at 1 month; Odds Ratio (OR) = 0.6909776, 95% CI 2-sided [0.4025454 to 1.1860776]
Statistical Analysis 2: Comparison: Team2BF vs Bright By Text; Test type: Superiority; p = 0.3, Cochran-Mantel-Haenszel — Value at 3 months; Odds Ratio (OR) = 0.6909776, 95% CI 2-sided [0.4025454 to 1.1860776]
Statistical Analysis 3: Comparison: Team2BF vs Bright By Text; Test type: Superiority; p = 0.3, Cochran-Mantel-Haenszel — Value at 6 months; Odds Ratio (OR) = 0.6909776, 95% CI 2-sided [0.4025454 to 1.1860776]

6. Secondary Outcome: Change in the Number of Participants Who Are Partially Breastfeeding as Measured by Participant Report/Chart Review
Time Frame: 1 month, 2 months, 3 months, 6 months postpartum
Population: A different number were analyzed at each time point
Measure: Count of Participants; unit: Participants
Arm/Group | Team2BF | Bright By Text
Number analyzed (Participants) | 35 | 37
Participants
  1 month postpartum: number analyzed (Participants) | 35 | 32
  1 month postpartum | 10 | 3
  2 months postpartum | 8 | 7
  3 months postpartum: number analyzed (Participants) | 35 | 36
  3 months postpartum | 7 | 4
  6 months postpartum: number analyzed (Participants) | 27 | 29
  6 months postpartum | 8 | 4
Statistical Analysis 1: Comparison: Team2BF vs Bright By Text; Test type: Superiority; p = 0.01692, Cochran-Mantel-Haenszel — Value at 1 month postpartum; Odds Ratio (OR) = 2.726859, 95% CI 2-sided [1.253958 to 5.929833]
Statistical Analysis 2: Comparison: Team2BF vs Bright By Text; Test type: Superiority; p = 0.7, Cochran-Mantel-Haenszel — Value at 2 months postpartum; Odds Ratio (OR) = 2.726859, 95% CI 2-sided [1.253958 to 5.929833]
Statistical Analysis 3: Comparison: Team2BF vs Bright By Text; Test type: Superiority; p = 0.3, Cochran-Mantel-Haenszel — Value at 3 months postpartum; Odds Ratio (OR) = 2.726859, 95% CI 2-sided [1.253958 to 5.929833]
Statistical Analysis 4: Comparison: Team2BF vs Bright By Text; Test type: Superiority; p = 0.15, Cochran-Mantel-Haenszel — Value at 6 months postpartum; Odds Ratio (OR) = 2.726859, 95% CI 2-sided [1.253958 to 5.929833]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Team2BF | Bright By Text
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT06375655/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/55/NCT06375655/ICF_001.pdf